CLINICAL TRIAL: NCT06598150
Title: Mapping Corticoreticulospinal Motor Control Using Brainstem and Spinal Cord fMRI in Chronic Hemiparetic Stroke
Brief Title: Mapping Corticoreticulospinal Motor Control in Chronic Hemiparetic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Molly Bright, Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00214855; 1R03HD113915-01 (NIH)
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Hemiparesis
Keywords: functional magnetic resonance imaging
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shoulder Abduction (Experimental)
  Interventions: Other: Shoulder Abduction

INTERVENTIONS:
Other: Shoulder Abduction — Individuals will be visually cued to perform short, unilateral, isometric shoulder abduction tasks. A visual display will provide real-time feedback of the shoulder abduction torque, to help the participant target a predetermined torque level.

SUMMARY:
This study uses functional magnetic resonance imaging to map neural activity throughout the central nervous system during a shoulder abduction task to characterize what motor pathways are being used post-stroke.

DETAILED DESCRIPTION:
Nearly 85% of stroke survivors experience significant unilateral impairment in upper extremity motor control, typically caused by damage to the corticospinal (CST) and corticoreticular (CRT) tracts (i.e., the corticofugal tracts). Alternative neural pathways, such as the contralesional cortico-reticulospinal tract (CRST), can be recruited to achieve movement of the affected arm and hand, but may have undesirable consequences. For example, the diffuse, bilateral branching of reticulospinal neurons can produce abnormal muscle co-activations (synergies) in the paretic limb, and involuntary mirror movements (associated reactions) between limbs. Together, these effects create stereotypical movement patterns post-stroke, and there is growing interest in novel "anti-synergy" interventions to enhance usage of residual CST systems rather than strengthening the CRST. Imaging has the potential to become an invaluable tool for evaluating whether rehabilitative strategies can preferentially access CST versus CRST pathways. However, current functional imaging research has focused on cortical activity, and must theoretically infer what pathway is used. Structural MRI directly assesses changes in white matter pathways, but it is limited to detecting long-term plasticity. To guide new interventions, there is a critical need to directly evaluate what descending motor pathways are active during movement. Thus, the overall objective of this study is to generate a novel fMRI dataset in participants with post-stroke hemiparesis, capturing neural activity during an innovative isometric shoulder abduction task, evaluating differences when abducting the paretic versus non-paretic arm. The investigators will acquire multi-echo fMRI data in individuals with post-stroke hemiparesis and age-matched controls, hypothesizing that increased reliance on the CRST will cause distinct activation patterns during shoulder abduction with the paretic limb, and that this will correlate with individual upper-extremity impairment (Upper-Extremity Fugl-Meyer Assessment). This work is significant because it will provide direct evidence of descending contralesional motor pathway involvement in post-stroke hemiparesis, and demonstrate the utility of neuroimaging for optimizing movements to preferentially engage specific systems and promote desired neural plasticity following injury.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged at least 18y
* Able to perform shoulder abduction task (confirmed during screening and initial examination)
* Safe to undergo MRI
* Able to follow visual instructions using MRI-compatible vision correction goggles
* No brainstem or cerebellar lesions
* No severe concurrent medical problems
* Cognitive/attentional capacity to focus on a task
* Able to communicate in English or Spanish

Additional inclusion criteria for stroke participants:

* Have sustained only one unilateral subcortical, ischemic lesion in the territory supplied by the Middle Cerebral Artery (confirmed by clinical or radiological reports) at least one year prior to participation in this project
* Paresis confined to one side, with moderate-to-severe motor impairment of the upper limb (Upper Extremity Fugl-Meyer score between 10 and 45).

Exclusion Criteria:

* MRI contraindications
* Severe claustrophobia
* Pregnant women
* Prisoners
* Vulnerable populations
* Diagnosis/history of:
* multiple sclerosis
* brain tumor
* brain radiation
* traumatic brain injury
* dementia
* Parkinson's disease
* Concurrent enrollment in an intervention study
* Concurrent use of medications known to suppress central nervous system activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
BOLD activation | 3 days to 3 months
  BOLD fMRI data will be analyzed to map neural activation associated with the shoulder abduction task.

CONTACTS AND LOCATIONS:
Overall Officials: Molly G Bright, DPhil, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
MR imaging data and the associated physiologic data collected during MRI scanning will be shared in an anonymized format. These data will be made available to public through the Open Science Framework (osf.io) or similar public repository. Code will be made available through the PI's laboratory Github account. A link to these resources will be included with publications resulting from this study to facilitate access.
Supporting Information: Analytic Code
Time Frame: At time of publication (or at project completion, whichever occurs first).
Access Criteria: Data will be anonymized and made publicly available, and at that time no approval is needed and therefore there are no access criteria.

DOCUMENTS (1):
  • Informed Consent Form (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT06598150/ICF_000.pdf